CLINICAL TRIAL: NCT00684112
Title: Analgesic Effects of Gabapentin After Scoliosis Surgery in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Arie Peliowski, Staff Anesthesiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1000010379
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Scoliosis
Keywords: pediatrics; Scoliosis; Gabapentin
MeSH Terms: conditions — Scoliosis | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Experimental): Single dose preoperative gabapentin
  Interventions: Drug: Gabapentin
- Placebo Control (Placebo Comparator): Single dose preoperative placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Patients in this arm of the study will receive two identical capsules, containing 300 mg of oral gabapentin each, 1 hour before surgery.
  Arms: Gabapentin
Drug: Placebo — Patients in this arm of the study will receive two identical placebo capsules 1 hour before surgery.
  Arms: Placebo Control

SUMMARY:
The primary aim of this study is to determine whether the use of gabapentin will improve postoperative analgesia and reduce opioid consumption and side effects in children undergoing corrective spinal surgery for idiopathic scoliosis. Secondary aims are to evaluate whether use of gabapentin reduces pain scores, decreases postoperative nausea and vomiting, decreases persisting pain and improves patient satisfaction.

DETAILED DESCRIPTION:
Surgical correction of scoliosis involves major orthopedic surgery, and can lead to severe acute postoperative pain and persistent neuropathic pain. The mainstays of treating postoperative pain are acetaminophen, non-steroidal anti-inflammatory drugs (NSAIDs), systemic opioids, and local anesthetic techniques. Despite being effective, their use is limited by adverse side effects. Acute postoperative pain involves multiple mechanisms and neural pathways, therefore a combination of different analgestic medications acting through different mechanisms, may be the most effective treatment. This strategy may also reduce the need for, and side effects of, using high doses of any one particular class of drugs.

Gabapentin is safe and well tolerated with few side effects and has minimal interactions with other drugs. The use of gabapentin to treat acute postoperative pain may improve quality of analgesia, result in decreased requirements for opioids and might consequently reduce the incidence of opioid induced side effects. It may also have a direct effect on postoperative nausea and vomiting, and decrease the incidence of persistent neuropathic pain. These qualities make gabapentin an attractive agent for use in management of postoperative pain in children undergoing corrective spinal injury.

The primary aim of this study is to determine whether the use of gabapentin will improve postoperative analgesia and reduce opioid consumption and side effects in children undergoing corrective spinal surgery for idiopathic scoliosis. Secondary aims are to evaluate whether use of gabapentin reduces pain scores, decreases postoperative nausea and vomiting, decreases persisting pain and improves patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 10 - 17 years of age
* scheduled for elective surgical correction of scoliosis
* able to operate a patient-controlled analgesia (PCA) pump

Exclusion Criteria:

* unable to cooperate
* unable to operate the PCA pump
* unable to rate pain
* have a known allergy or sensitivity to gabapentin or morphine
* have a history of chronic pain or daily analgesic use
* have taken acetaminophen, a non-steroidal anti-inflammatory drug, or an antacid within a 24-hour period prior to surgery

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption postoperatively. | 0 to 24 hours postoperatively

SECONDARY OUTCOMES:
Time to first rescue analgesia. | Determined by outcome
Pain intensity scores at rest and with movement | Assessed at 1 hour, 4 hours, 12 hours, 24 hours, 72 hours, and 1 week postoperatively and at the 6-week outpatient follow up visit.
Incidence and severity of nausea, vomiting, pruritis, sedation, dizziness, and presence of persisting pain symptoms | Assessed at 1 hour, 4 hours, 12 hours, 24 hours, and 48 hours postoperatively.
Time to first postoperative oral intake as a measure of bowel function. | Determined by outcome

CONTACTS AND LOCATIONS:
Overall Officials: Arie Peliowski, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada